CLINICAL TRIAL: NCT03307252
Title: The Effect of Potent Inhibitors of Drug Transporters (Verapamil, Rifampin, Cimetidine, Probenecid) on Pharmacokinetics of a Transporter Probe Drug Cocktail Consisting of Digoxin, Furosemide, Metformin and Rosuvastatin (an Open-label, Randomised, Crossover Trial in Three Parts)
Brief Title: This Study Tests the Effect of Certain Medicines on the Transport of Other Medicines in the Body of Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 0352-2100; 2017-001549-29 (EudraCT Number)
Record Dates: First submitted 2017-10-06; First posted 2017-10-11 (Actual); Results first posted 2019-07-12 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Healthy
MeSH Terms: interventions — Digoxin; Furosemide; Metformin; Rosuvastatin Calcium; Verapamil; Rifampin; Cimetidine; Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Treatment Reference 1 (Experimental)
  Interventions: Drug: Digoxin; Drug: Furosemide; Drug: Metformin; Drug: Rosuvastatin
- Treatment Reference 2 (Experimental)
  Interventions: Drug: Metformin
- Treatment Reference 3 (Experimental)
  Interventions: Drug: Furosemide
- Treatment 1 (Experimental)
  Interventions: Drug: Digoxin; Drug: Furosemide; Drug: Metformin; Drug: Rosuvastatin; Drug: Verapamil
- Treatment 2 (Experimental)
  Interventions: Drug: Digoxin; Drug: Furosemide; Drug: Metformin; Drug: Rosuvastatin; Drug: Rifampin
- Treatment 3 (Experimental)
  Interventions: Drug: Digoxin; Drug: Furosemide; Drug: Metformin; Drug: Rosuvastatin; Drug: Cimetidine
- Treatment 4 (Experimental)
  Interventions: Drug: Digoxin; Drug: Furosemide; Drug: Metformin; Drug: Rosuvastatin; Drug: Probenecid
- Treatment 5 (Experimental)
  Interventions: Drug: Metformin; Drug: Cimetidine
- Treatment 6 (Experimental)
  Interventions: Drug: Furosemide; Drug: Probenecid

INTERVENTIONS:
Drug: Digoxin — Tablet
  Arms: Treatment 1; Treatment 2; Treatment 3; Treatment 4; Treatment Reference 1
Drug: Furosemide — Oral solution
  Arms: Treatment 1; Treatment 2; Treatment 3; Treatment 4; Treatment 6; Treatment Reference 1; Treatment Reference 3
Drug: Metformin — Oral solution
  Arms: Treatment 1; Treatment 2; Treatment 3; Treatment 4; Treatment 5; Treatment Reference 1; Treatment Reference 2
Drug: Rosuvastatin — Film-coated tablet
  Arms: Treatment 1; Treatment 2; Treatment 3; Treatment 4; Treatment Reference 1
Drug: Verapamil — Film-coated tablet
  Arms: Treatment 1
Drug: Rifampin — Film-coated tablet
  Arms: Treatment 2
Drug: Cimetidine — Tablet
  Arms: Treatment 3; Treatment 5
Drug: Probenecid — Tablet
  Arms: Treatment 4; Treatment 6

SUMMARY:
The primary objective of this trial is to investigate the relative bioavailabilities of digoxin, furosemide, metformin and rosuvastatin given as a cocktail alone and as a cocktail together with the following drug transporter inhibitors:

Part 1: verapamil (P-gp) and rifampin (OATP1B1/1B3) Part 2: cimetidine (OCT2/MATE) Part 3: probenecid (OAT1/3) The secondary objective is to investigate other potential changes in pharmacokinetics (e.g. in clearance, volume of distribution, etc.) of digoxin, furosemide, metformin and rosuvastatin given as a cocktail alone and as a cocktail together with the inhibitors describe above.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients, sulphonamides, or cardiac glycosides)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 24 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Male subjects with Women of child bearing potential (WOCBP) partner who are unwilling to use male contraception (condom or sexual abstinence) from the first administration of trial medication until 30 days after last administration of trial medication
* Hypokalemia, hypomagnesemia, or hypercalcemia
* PQ interval greater than 220 ms in the Electrocardiogram (ECG) at screening
* Marked conductivity disorders (e.g. sinu-atrial blocks of II° or III°)
* Myopathy
* Hereditary galactose or fructose intolerance, lactase deficiency, or glucose-galactose malabsorption
* History of nephrolithiasis
* Gout or clinically relevant elevation of uric acid
* Creatinine clearance (according to CKD EPI formula) is lower than 80 ml/min
* Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CTC North GmbH & Co. KG, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial consisted of 3 parts investigating different drug transporter inhibitors. All parts of the trial were performed in healthy male participants in a randomised, open-label, three-way (Part 1) or four-way (Part 2 and 3) crossover design.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants were not to be randomised to trial treatment if any of the in- or exclusion criteria were violated at screening.
Groups:
- Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1): In trial part 1 participants were administered a single dose of Cocktail (reference treatment 1, R1) with 280 milliliter (mL) of water in period 1. R1 is a drug cocktail that contains a single dose of each, 0.25 milligram (mg) Digoxin tablet, 1 mg Furosemide oral solution, 10 mg Metformin oral solution and 10 mg Rosuvastatin film-coated tablet. Followed by a single dose of 120 mg Verapamil orally with 240 mL of water at 1 hour (h) prior to R1 which is administered with 280 mL of water in period 2. In period 3 participants were administered a single dose of 600 mg Rifampin film-coated tablet with 280 mL of water together with R1. Treatment periods were separated by a wash-out period of 13 days.
- (Verapamil + R1)/ (Rifampin + R1)/ R1: In trial part 1 participants were administered a single dose of 120 mg Verapamil orally with 240 mL of water at 1 h prior to R1 which is administered with 280 mL of water in period 1. Followed by a single dose of 600 mg Rifampin film-coated tablet orally with 280 mL of water together with R1 in period 2. In period 3 participants were administered a single dose of R1 with 280 milliliter (mL) of water. R1 is a drug cocktail that contains a single dose of each, 0.25 milligram (mg) Digoxin tablet, 1 mg Furosemide oral solution, 10 mg Metformin oral solution and 10 mg Rosuvastatin film-coated tablet. Treatment periods were separated by a wash-out period of 13 days.
- (Rifampin + R1)/ R1/ (Verapamil + R1): In trial part 1 participants were administered a single dose of 600 mg Rifampin film-coated tablet orally with 280 mL of water together with R1 in period 1. Followed by a single dose of R1 with 280 mL of water in period 2. R1 is a drug cocktail that contains a single dose of each, 0.25 mg Digoxin tablet, 1 mg Furosemide oral solution, 10 mg Metformin oral solution and 10 mg Rosuvastatin film-coated tablet. In period 3 participants were administered a single dose of 120 mg Verapamil orally with 240 mL of water at 1 hour (h) prior to the R1 which is administered with 280 mL of water. Treatment periods were separated by a wash-out period of 13 days.
- R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin): In trial part 2 participants were administered single dose of R1 which is administered with 280 mL of water in period 1. R1 is a drug cocktail that contains a single dose of each 0.25 milligram (mg) Digoxin tablet, 1 mg Furosemide oral solution, 10 mg Metformin oral solution and 10 mg Rosuvastatin film-coated tablet. Followed by single therapeutic dose of 500 mg Metformin oral solution with 280 mL of water in period 2. Followed by 400 mg Cimetidine 1 orally at 1 h prior to R1 and at 4 h, 8 h, 12 h, 24 h (Day 2) and 36 h after R1 (Day 2) in period 3. Followed by 400 mg Cimetidine 1 tablet orally at 1 h prior to therapeutic dose of 500mg of Metformin and at 4 h, 8 h, 12, 24 h (Day 2) and 36 h after metformin (Day 2) in period 4. All doses of Cimetidine administered with 240 mL water and R1 and dose of Metformin with 280 mL of water. Treatment periods were separated by a wash-out period of at least 7 days.
- Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1): In trial part 2 participants were administered single therapeutic dose of 500 mg Metformin oral solution with 280 mL of water in period 1. Followed by 400 mg Cimetidine 1 tablet orally at 1 h prior to Metformin and at 4 h, 8 h, 12, 24 h (Day 2) and 36 h after metformin (Day 2) in period 2. Followed by a single dose of R1 with 280 mL of water in period 3. R1 is a drug cocktail that contains single dose of each 0.25 milligram (mg) Digoxin tablet, 1 mg Furosemide oral solution, 10 mg Metformin oral solution and 10 mg Rosuvastatin film-coated tablet. Followed by 400 mg Cimetidine 1 orally at 1 h prior to R1 and at 4 h, 8 h, 12 h, 24 h (Day 2) and 36 h after R1 (Day 2) in period 4. All doses of Cimetidine administered with 240 mL water and R1 and dose of Metformin with 280 mL of water. Treatment periods were separated by a wash-out period of at least 7 days.
- (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin: In trial part 2 participants were administered 400 mg Cimetidine 1 tablet orally at 1 h prior to R1 and at 4 h, 8 h, 12 h, 24 h (Day 2) and 36 h after R1 (Day 2) in period 1. Followed by single dose of R1 which is administered with 280 mL of water in period 1. R1 is a drug cocktail that contains single dose of each 0.25 mg Digoxin tablet, 1 mg Furosemide oral solution, 10 mg Metformin oral solution and 10 mg Rosuvastatin film-coated tablet in period 2. Followed by 400 mg Cimetidine 1 tablet orally at 1 h prior to Metformin and at 4 h, 8 h, 12, 24 h (Day 2) and 36 h after Metformin (Day 2) in period 3. Followed by single therapeutic dose of 500 mg Metformin oral solution with 280 mL of water in period 4. All doses of Cimetidine administered with 240 mL water and R1 and dose of Metformin with 280 mL of water. Treatment periods were separated by a wash-out period of at least 7 days.
- (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1: In trial part 2 participants were administered 400 mg Cimetidine 1 tablet orally at 1 h prior to Metformin and at 4 h, 8 h, 12, 24 h (Day 2) and 36 h after Metformin (Day 2) in period 1. Followed by 400 mg Cimetidine 1 tablet orally at 1 h prior to R1 and at 4 h, 8 h, 12 h, 24 h (Day 2) and 36 h after R1 (Day 2) in period 2. Followed by single therapeutic dose of 500 mg Metformin oral solution with 280 mL of water in period 3. Followed by single dose of R1 which is administered with 280 mL of water in period 1. R1 is a drug cocktail that contains single dose of each 0.25 mg Digoxin tablet, 1 mg Furosemide oral solution, 10 mg Metformin oral solution and 10 mg Rosuvastatin film-coated tablet in period 4. All doses of Cimetidine administered with 240 mL water and R1 and dose of Metformin with 280 mL of water. Treatment periods were separated by a wash-out period of at least 7 days.
- R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide): In trial part 3 participants were administered single dose of R1 which is administered with 280 mL of water in period 1. R1 is a drug cocktail that contains single dose of each 0.25 mg Digoxin tablet, 1 mg Furosemide oral solution, 10 mg Metformin oral solution and 10 mg Rosuvastatin film-coated tablet. Followed by single therapeutic dose of 40 mg Furosemide oral solution with 280 mL of water in period 2. Followed by 2 tablets of 500 mg Probenecid (2*500 mg) administered orally 13 h prior and again 1 h prior to the administration of R1 on day 1 in period 3. Followed by 2 tablets of 500 mg Probenecid (2*500 mg) administered orally 13 hours prior and again 1 h prior to the administration of Furosemide on Day 1 in period 4. All doses of Cimetidine administered with 240 mL water and dose of Furosemide and R1 with 280 mL of water. Treatment periods were separated by a wash-out period of at least 7 days.
- Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1): In trial part 3 participants were administered single therapeutic dose of 40 mg Furosemide oral solution with 280 mL of water in period 1. Followed by 2 tablets of 500 mg Probenecid (2*500 mg) administered orally 13 hours prior and again 1 h prior to the administration of Furosemide on Day 1 in period 2. Followed by single dose of R1 which is administered with 280 milliliter (mL) of water in period 3. R1 is a drug cocktail that contains single dose of each 0.25 milligram (mg) Digoxin tablet, 1 mg Furosemide oral solution, 10 mg Metformin oral solution and 10 mg Rosuvastatin film-coated tablet. Followed by 2 tablets of 500 mg Probenecid (2*500 mg) administered orally 13 h prior and again 1 h prior to the administration of R1 on day 1 in period 4. All doses of Cimetidine administered with 240 mL water and dose of Furosemide and R1 with 280 mL of water. Treatment periods were separated by a wash-out period of at least 7 days.
- (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide: In trial part 3 participants were administered 2 tablets of 500 mg Probenecid (2*500 mg) administered orally 13 h prior and again 1 h prior to the administration of R1 on day 1 in period 1. Followed by single dose of R1 which is administered with 280 mL of water in period 2. R1 is a drug cocktail that contains single dose of each 0.25 mg Digoxin tablet, 1 mg Furosemide oral solution, 10 mg Metformin oral solution and 10 mg Rosuvastatin film-coated tablet. Followed by 2 tablets of 500 mg Probenecid (2*500 mg) administered orally 13 hours prior and again 1 h prior to the administration of Furosemide on Day 1 in period 3. Followed by single therapeutic dose of 40 mg Furosemide oral solution with 280 mL of water in period 4. All doses of Cimetidine administered with 240 mL water and dose of Furosemide and R1 with 280 mL of water. Treatment periods were separated by a wash-out period of at least 7 days.
- (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1: In trial part 3 participants were administered 2 tablets of 500 mg Probenecid (2*500 mg) administered orally 13 hours prior and again 1 h prior to the administration of Furosemide on Day 1 in period 1. Followed by 2 tablets of 500 mg Probenecid (2*500 mg) administered orally 13 h prior and again 1 h prior to the administration of R1 on day 1 in period 2. Followed by single therapeutic dose of 40 mg Furosemide oral solution with 280 mL of water in period 3. Followed by single dose of R1 which is administered with 280 milliliter (mL) of water in period 4. R1 is a drug cocktail that contains a single dose of each 0.25 milligram (mg) Digoxin tablet, 1 mg Furosemide oral solution, 10 mg Metformin oral solution and 10 mg Rosuvastatin film-coated tablet. All doses of Cimetidine administered with 240 mL water and dose of Furosemide and R1 with 280 mL of water. Treatment periods were separated by a wash-out period of at least 7 days.
Period: Part 1, Period 1
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 4 (Participants randomised in Part 1) | 4 (Participants randomised in Part 1) | 4 (Participants randomised in Part 1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1, Washout Period 1 (13 Days)
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1, Period 2
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 4 (Participants randomised in Part 1) | 4 (Participants randomised in Part 1) | 4 (Participants randomised in Part 1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1, Washout Period 2 (13 Days)
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1, Period 3
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 4 (Participants randomised in Part 1) | 4 (Participants randomised in Part 1) | 4 (Participants randomised in Part 1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2, Period 1
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 0 | 0 | 0 | 4 (Participants randomized in Part 2) | 4 (Participants randomized in Part 2) | 4 (Participants randomized in Part 2) | 5 (Participants randomized in Part 2) | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 4 | 4 | 3 | 5 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Treatment not received | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 2, Washout Period 1 (7 Days)
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 0 | 0 | 0 | 4 | 4 | 3 | 5 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 4 | 4 | 3 | 5 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2, Period 2
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 0 | 0 | 0 | 4 | 4 | 3 | 5 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 4 | 4 | 3 | 5 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2, Washout Period 2 (7 Days)
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 0 | 0 | 0 | 4 | 4 | 3 | 5 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 4 | 4 | 3 | 5 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2, Period 3
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 0 | 0 | 0 | 4 | 4 | 3 | 5 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 4 | 3 | 3 | 5 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other than listed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2, Washout Period 3 (7 Days)
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 0 | 0 | 0 | 4 | 3 | 3 | 5 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 4 | 3 | 3 | 4 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Part 2, Period 4
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 0 | 0 | 0 | 4 | 3 | 3 | 5 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 4 | 3 | 3 | 4 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other than listed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Part 3, Period 1
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 (Participants randomized in Part 3) | 4 (Participants randomized in Part 3) | 4 (Participants randomized in Part 3) | 4 (Participants randomized in Part 3)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3, Washout Period 1 (7 Days)
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3, Period 2
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3, Washout Period 2 (7 Days)
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3, Period 3
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3, Washout Period 3 (7 Days)
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Treatment not received due to AE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Part 3, Period 4
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All subjects who were dispended study medication and were documented to have taken at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cocktail (R1)/ (Verapamil + R1)/ (Rifampin + R1) | (Verapamil + R1)/ (Rifampin + R1)/ R1 | (Rifampin + R1)/ R1/ (Verapamil + R1) | R1/ Metformin/ (Cimetidine+R1)/ (Cimetidine+Metformin) | Metformin/ (Cimetidine+Metformin)/ R1/ (Cimetidine+R1) | (Cimetidine+R1)/ R1/ (Cimetidine+Metformin)/ Metformin | (Cimetidine+Metformin)/ (Cimetidine+R1)/ Metformin/ R1 | R1/ Furosemide/ (Probenecid + R1)/ (Probenecid + Furosemide) | Furosemide/ (Probenecid + Furosemide)/ R1/ (Probenecid + R1) | (Probenecid + R1)/ R1/ (Probenecid + Furosemide)/ Furosemide | (Probenecid + Furosemide)/ (Probenecid + R1)/ Furosemide/ R1 | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 5 | 4 | 4 | 4 | 4 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Part 1 | 30.0 (6.8) | 51.5 (1.3) | 36.3 (10.6) | 32.8 (10.2) | 38.3 (13.1) | 35.3 (11.1) | 41.6 (10.5) | 29.3 (7.9) | 30.0 (8.8) | 33.0 (13.2) | 43.5 (8.1) | 36.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 4 | 4 | 4 | 4 | 4 | 4 | 5 | 4 | 4 | 4 | 4 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 4 | 4 | 4 | 4 | 5 | 4 | 4 | 4 | 4 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 4 | 4 | 4 | 4 | 3 | 5 | 4 | 4 | 4 | 4 | 44
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz) (Verapamil + R1 (T1) vs. R1)
Description: AUC0-tz, area under the concentration-time curve of the analytes: digoxin, furosemide, metformin, and rosuvastatin (at cocktail doses) in plasma over the time interval from 0 to the last quantifiable data point is presented. Geometric mean (gMean) presented here is an adjusted gMean and standard error (SE) presented is a geometric SE (gSE).
Time Frame: Samples were taken within 0:20 hour:minutes (hh:mm) prior to first study drug administration and at 0:20, 0:40, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 8:00, 10:00, 11:00, 12:00, 24:00, 36:00, 47:00, 71:00 and 95:00 after drug administration.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): All subjects in the TS providing at least 1 primary or secondary PK parameter that was not excluded due to a protocol violation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Standard Error); unit: Nanomole*hour/litre (nmol*h/L)
Groups:
- Verapamil + R1 (T1): Participants were administered a single dose of 120 mg Verapamil orally with 240 mL of water at 1 h prior to the R1 which is administered with 280 mL of water in trial part 1.
- Cocktail (R1): Participants were administered a single dose of Cocktail (reference treatment 1, R1) with 280 mL of water. R1 is a drug cocktail that contains a single dose of each, 0.25 mg Digoxin tablet, 1 mg Furosemide oral solution, 10 mg Metformin oral solution and 10 mg Rosuvastatin film-coated tablet in trial part 1, 2 and 3.
Arm/Group | Verapamil + R1 (T1) | Cocktail (R1)
Number analyzed (Participants) | 12 | 12
Nanomole*hour/litre (nmol*h/L)
  Digoxin | 13.71 (1.10) | 13.61 (1.10)
  Furosemide | 165.80 (1.06) | 176.85 (1.06)
  Metformin | 1126.22 (1.05) | 1357.34 (1.05)
  Rosuvastatin | 98.98 (1.11) | 87.29 (1.11)
Statistical Analysis 1: Comparison: Verapamil + R1 (T1) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted geometric mean (gMean) ratio = 100.70, 90% CI 2-sided [88.84 to 114.15], Standard Error of Mean 17.9 — Standard Error of the mean is actually intra individual geometric coefficient of variation (gCV). Adjusted gMean ratio is given for T1 vs. R1; Digoxin, Analysis of variance (ANOVA) model on the logarithmic scale includes effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed
Statistical Analysis 2: Comparison: Verapamil + R1 (T1) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean ratio = 93.76, 90% CI 2-sided [86.12 to 102.06], Standard Error of Mean 12.1 — [estimate comment as in outcome 1, analysis 1]; Furosemide, ANOVA model on the logarithmic scale includes effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed
Statistical Analysis 3: Comparison: Verapamil + R1 (T1) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 82.97, 90% CI 2-sided [76.96 to 89.46], Standard Error of Mean 10.7 — [estimate comment as in outcome 1, analysis 1]; Metformin, ANOVA model on the logarithmic scale includes effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed
Statistical Analysis 4: Comparison: Verapamil + R1 (T1) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 113.40, 90% CI 2-sided [97.62 to 131.72], Standard Error of Mean 21.5 — [estimate comment as in outcome 1, analysis 1]; Rosuvastatin, ANOVA model on the logarithmic scale includes effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed

2. Primary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz) (Rifampin + R1 (T2) vs. R1)
Description: AUC0-tz, area under the concentration-time curve of the analytes: digoxin, furosemide, metformin, and rosuvastatin (at cocktail doses) in plasma over the time interval from 0 to the last quantifiable data point is presented. gMean presented here is an adjusted gMean and SE presented is a gSE.
Time Frame: Samples were taken within 0:20 hh:mm prior to first study drug administration and at 0:20, 0:40, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 8:00, 10:00, 11:00, 12:00, 24:00, 36:00, 47:00, 71:00 and 95:00 after drug administration.
Population: PKS
Measure: Geometric Mean (Standard Error); unit: Nanomole*hour/litre (nmol*h/L)
Groups:
- Rifampin + R1 (T2): Participants were administered a single dose of 600 mg Rifampin film-coated tablet orally with 280 mL of water together with Cocktail in trial part 1.
Arm/Group | Rifampin + R1 (T2) | Cocktail (R1)
Number analyzed (Participants) | 12 | 12
Nanomole*hour/litre (nmol*h/L)
  Digoxin | 17.89 (1.10) | 13.61 (1.10)
  Furosemide | 211.82 (1.06) | 176.85 (1.06)
  Metformin | 1473.38 (1.05) | 1357.34 (1.05)
  Rosuvastatin | 303.81 (1.11) | 87.29 (1.11)
Statistical Analysis 1: Comparison: Rifampin + R1 (T2) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted geometric mean (gMean) ratio = 131.41, 90% CI 2-sided [115.93 to 148.97], Standard Error of Mean 17.9 — Standard Error of the mean is actually intra individual geometric coefficient of variation (gCV). Adjusted gMean ratio is given for T2 vs. R1; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Rifampin + R1 (T2) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean ratio = 119.78, 90% CI 2-sided [110.03 to 130.39], Standard Error of Mean 12.1 — [estimate comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Rifampin + R1 (T2) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 108.55, 90% CI 2-sided [100.68 to 117.03], Standard Error of Mean 10.7 — [estimate comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Rifampin + R1 (T2) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 348.06, 90% CI 2-sided [299.64 to 404.31], Standard Error of Mean 21.5 — [estimate comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 4]

3. Primary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz) (Cimetidine + R1 (T3) vs. R1)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Standard Error); unit: Nanomole*hour/litre (nmol*h/L)
Groups:
- Cimetidine + R1 (T3): Participants were administered 400 mg Cimetidine 1 tablet orally at 1 h prior to cocktail and at 4 h, 8 h, 12 h, 24 h (Day 2) and 36 h after cocktail (Day 2). All doses of Cimetidine administered with 240 mL water and dose of Cocktail with 280 mL of water in trial part 2.
Arm/Group | Cimetidine + R1 (T3) | Cocktail (R1)
Number analyzed (Participants) | 15 | 13
Nanomole*hour/litre (nmol*h/L)
  Digoxin | 19.03 (1.07) | 15.15 (1.07)
  Furosemide | 196.39 (1.05) | 194.05 (1.05)
  Metformin | 2006.60 (1.06) | 1532.41 (1.07)
  Rosuvastatin | 139.54 (1.13) | 129.90 (1.13)
Statistical Analysis 1: Comparison: Cimetidine + R1 (T3) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted geometric mean (gMean) ratio = 125.61, 90% CI 2-sided [113.99 to 138.43], Standard Error of Mean 13.2 — Standard Error of the mean is actually intra individual geometric coefficient of variation (gCV). Adjusted gMean ratio is given for T3 vs. R1; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cimetidine + R1 (T3) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean ratio = 101.21, 90% CI 2-sided [94.59 to 108.30], Standard Error of Mean 9.2 — [estimate comment as in outcome 3, analysis 1]; [other analysis details as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cimetidine + R1 (T3) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 130.94, 90% CI 2-sided [119.82 to 143.10], Standard Error of Mean 13.6 — [estimate comment as in outcome 3, analysis 1]; [other analysis details as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Cimetidine + R1 (T3) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 107.42, 90% CI 2-sided [97.57 to 118.27], Standard Error of Mean 12.9 — [estimate comment as in outcome 3, analysis 1]; [other analysis details as in outcome 1, analysis 4]

4. Primary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz) (Probenecid + R1 (T4) vs. R1)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Standard Error); unit: Nanomole*hour/litre (nmol*h/L)
Groups:
- Probenecid + R1 (T4): Participants were administered 2 tablets of 500 mg Probenecid (2*500 mg) orally 13 h prior and again 1 h prior to the administration of R1 on day 1. All doses of Cimetidine administered with 240 mL water and dose of R1 which is administered with 280 mL of water in trial part 3.
Arm/Group | Probenecid + R1 (T4) | Cocktail (R1)
Number analyzed (Participants) | 15 | 16
Nanomole*hour/litre (nmol*h/L)
  Digoxin | 14.44 (1.08) | 13.52 (1.08)
  Furosemide | 483.38 (1.08) | 177.96 (1.07)
  Metformin | 1331.83 (1.08) | 1321.20 (1.08)
  Rosuvastatin | 238.16 (1.10) | 106.69 (1.10)
Statistical Analysis 1: Comparison: Probenecid + R1 (T4) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted geometric mean (gMean) ratio = 106.78, 90% CI 2-sided [96.51 to 118.15], Standard Error of Mean 15.5 — Standard Error of the mean is actually intra individual geometric coefficient of variation (gCV). Adjusted gMean ratio is given for T4 vs. R1; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Probenecid + R1 (T4) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean ratio = 271.63, 90% CI 2-sided [246.74 to 299.03], Standard Error of Mean 15.9 — [estimate comment as in outcome 4, analysis 1]; [other analysis details as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Probenecid + R1 (T4) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 100.80, 90% CI 2-sided [94.62 to 107.39], Standard Error of Mean 9.6 — [estimate comment as in outcome 4, analysis 1]; [other analysis details as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Probenecid + R1 (T4) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 223.24, 90% CI 2-sided [203.79 to 244.55], Standard Error of Mean 13.9 — [estimate comment as in outcome 4, analysis 1]; [other analysis details as in outcome 1, analysis 4]

5. Primary Outcome: Maximum Measured Concentration of the Analytes: Digoxin, Furosemide, Metformin, and Rosuvastatin (Cmax) (T1 vs. R1)
Description: Cmax, maximum measured concentration of the analytes: digoxin, furosemide, metformin, and rosuvastatin (at cocktail doses) is presented. gMean presented here is an adjusted gMean and SE presented is a gSE.
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Standard Error); unit: Nanomole/ litre (nmol/ L)
Arm/Group | Verapamil + R1 (T1) | Cocktail (R1)
Number analyzed (Participants) | 12 | 12
Nanomole/ litre (nmol/ L)
  Digoxin | 1.42 (1.09) | 1.17 (1.09)
  Furosemide | 84.32 (1.06) | 88.59 (1.06)
  Metformin | 179.45 (1.04) | 223.78 (1.04)
  Rosuvastatin | 7.90 (1.14) | 6.84 (1.14)
Statistical Analysis 1: Comparison: Verapamil + R1 (T1) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted geometric mean (gMean) ratio = 121.64, 90% CI 2-sided [100.43 to 147.33], Standard Error of Mean 27.7 — [estimate comment as in outcome 1, analysis 1]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Verapamil + R1 (T1) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean ratio = 95.18, 90% CI 2-sided [83.03 to 109.11], Standard Error of Mean 19.6 — [estimate comment as in outcome 1, analysis 1]; [other analysis details as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Verapamil + R1 (T1) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 80.19, 90% CI 2-sided [73.01 to 88.08], Standard Error of Mean 13.4 — [estimate comment as in outcome 1, analysis 1]; [other analysis details as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Verapamil + R1 (T1) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 115.39, 90% CI 2-sided [93.80 to 141.94], Standard Error of Mean 30.1 — [estimate comment as in outcome 1, analysis 1]; [other analysis details as in outcome 1, analysis 4]

6. Primary Outcome: Maximum Measured Concentration of the Analytes: Digoxin, Furosemide, Metformin, and Rosuvastatin (Cmax) (T2 vs. R1)
Description: as for outcome 5
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Standard Error); unit: Nanomole/ litre (nmol/ L)
Arm/Group | Rifampin + R1 (T2) | Cocktail (R1)
Number analyzed (Participants) | 12 | 12
Nanomole/ litre (nmol/ L)
  Digoxin | 2.55 (1.09) | 1.17 (1.09)
  Furosemide | 119.66 (1.06) | 88.59 (1.06)
  Metformin | 251.32 (1.04) | 223.78 (1.04)
  Rosuvastatin | 77.00 (1.14) | 6.84 (1.14)
Statistical Analysis 1: Comparison: Rifampin + R1 (T2) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted geometric mean (gMean) ratio = 218.26, 90% CI 2-sided [180.19 to 264.36], Standard Error of Mean 27.7 — [estimate comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Rifampin + R1 (T2) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean ratio = 135.07, 90% CI 2-sided [117.83 to 154.84], Standard Error of Mean 19.6 — [estimate comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Rifampin + R1 (T2) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 112.31, 90% CI 2-sided [102.26 to 123.35], Standard Error of Mean 13.4 — [estimate comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Rifampin + R1 (T2) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 1125.10, 90% CI 2-sided [914.63 to 1384.00], Standard Error of Mean 30.1 — [estimate comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 4]

7. Primary Outcome: Maximum Measured Concentration of the Analytes: Digoxin, Furosemide, Metformin, and Rosuvastatin (Cmax) (T3 vs. R1)
Description: as for outcome 5
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Standard Error); unit: Nanomole/ litre (nmol/ L)
Arm/Group | Cimetidine + R1 (T3) | Cocktail (R1)
Number analyzed (Participants) | 15 | 13
Nanomole/ litre (nmol/ L)
  Digoxin | 1.65 (1.07) | 1.35 (1.08)
  Furosemide | 97.69 (1.08) | 93.23 (1.08)
  Metformin | 316.83 (1.07) | 258.33 (1.08)
  Rosuvastatin | 13.21 (1.15) | 11.30 (1.15)
Statistical Analysis 1: Comparison: Cimetidine + R1 (T3) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted geometric mean (gMean) ratio = 218.26, 90% CI 2-sided [180.19 to 264.36], Standard Error of Mean 27.7 — [estimate comment as in outcome 3, analysis 1]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cimetidine + R1 (T3) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean ratio = 104.78, 90% CI 2-sided [89.97 to 122.03], Standard Error of Mean 21.0 — [estimate comment as in outcome 3, analysis 1]; [other analysis details as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cimetidine + R1 (T3) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 122.65, 90% CI 2-sided [107.68 to 139.69], Standard Error of Mean 20.1 — [estimate comment as in outcome 4, analysis 1]; [other analysis details as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Cimetidine + R1 (T3) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 116.88, 90% CI 2-sided [105.07 to 130.03], Standard Error of Mean 14.4 — [estimate comment as in outcome 3, analysis 1]; [other analysis details as in outcome 1, analysis 4]

8. Primary Outcome: Maximum Measured Concentration of the Analytes: Digoxin, Furosemide, Metformin, and Rosuvastatin (Cmax) (T4 vs. R1)
Description: as for outcome 5
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Standard Error); unit: Nanomole/ litre (nmol/ L)
Arm/Group | Probenecid + R1 (T4) | Cocktail (R1)
Number analyzed (Participants) | 15 | 16
Nanomole/ litre (nmol/ L)
  Digoxin | 1.13 (1.07) | 1.30 (1.07)
  Furosemide | 110.64 (1.07) | 90.00 (1.07)
  Metformin | 246.78 (1.12) | 243.49 (1.12)
  Rosuvastatin | 43.29 (1.11) | 10.11 (1.10)
Statistical Analysis 1: Comparison: Probenecid + R1 (T4) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted geometric mean (gMean) ratio = 87.07, 90% CI 2-sided [76.08 to 99.64], Standard Error of Mean 20.9 — [estimate comment as in outcome 4, analysis 1]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Probenecid + R1 (T4) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean ratio = 122.94, 90% CI 2-sided [110.25 to 137.09], Standard Error of Mean 18.0 — [estimate comment as in outcome 4, analysis 1]; [other analysis details as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Probenecid + R1 (T4) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 101.35, 90% CI 2-sided [93.65 to 109.70], Standard Error of Mean 12.0 — [estimate comment as in outcome 4, analysis 1]; [other analysis details as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Probenecid + R1 (T4) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 428.23, 90% CI 2-sided [359.78 to 509.70], Standard Error of Mean 26.8 — [estimate comment as in outcome 4, analysis 1]; [other analysis details as in outcome 1, analysis 4]

9. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞) (T1 vs. R1)
Description: AUC0-∞, area under the concentration-time curve of the analytes: digoxin, furosemide, metformin, and rosuvastatin (at cocktail doses) in plasma over the time interval from 0 extrapolated to infinity is presented. AUC0-∞ not displayed for Digoxin analyte as precision was considered non-sufficient. gMean presented here is an adjusted gMean and SE presented is a gSE.
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Standard Error); unit: Nanomole*hour/litre (nmol*h/L)
Arm/Group | Verapamil + R1 (T1) | Cocktail (R1)
Number analyzed (Participants) | 12 | 12
Nanomole*hour/litre (nmol*h/L)
  Furosemide | 176.44 (1.06) | 191.29 (1.06)
  Metformin | 1147.23 (1.05) | 1365.85 (1.05)
  Rosuvastatin | 116.80 (1.10) | 94.14 (1.10)
Statistical Analysis 1: Comparison: Verapamil + R1 (T1) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean ratio = 92.24, 90% CI 2-sided [85.28 to 99.76], Standard Error of Mean 11.2 — [estimate comment as in outcome 1, analysis 1]; [other analysis details as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Verapamil + R1 (T1) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 83.99, 90% CI 2-sided [78.32 to 90.08], Standard Error of Mean 10.0 — [estimate comment as in outcome 1, analysis 1]; [other analysis details as in outcome 1, analysis 3]
Statistical Analysis 3: Comparison: Verapamil + R1 (T1) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 124.06, 90% CI 2-sided [105.11 to 146.43], Standard Error of Mean 23.9 — [estimate comment as in outcome 1, analysis 1]; [other analysis details as in outcome 1, analysis 4]

10. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞) (T2 vs. R1)
Description: as for outcome 9
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Standard Error); unit: Nanomole*hour/litre (nmol*h/L)
Arm/Group | Rifampin + R1 (T2) | Cocktail (R1)
Number analyzed (Participants) | 12 | 12
Nanomole*hour/litre (nmol*h/L)
  Furosemide | 215.63 (1.06) | 191.29 (1.06)
  Metformin | 1482.76 (1.05) | 1365.85 (1.05)
  Rosuvastatin | 320.72 (1.10) | 94.14 (1.10)
Statistical Analysis 1: Comparison: Rifampin + R1 (T2) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 112.73, 90% CI 2-sided [104.23 to 121.92], Standard Error of Mean 11.2 — [estimate comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Rifampin + R1 (T2) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 108.56, 90% CI 2-sided [101.22 to 116.43], Standard Error of Mean 10.0 — [estimate comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 3]
Statistical Analysis 3: Comparison: Rifampin + R1 (T2) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 340.67, 90% CI 2-sided [288.63 to 402.10], Standard Error of Mean 23.9 — [estimate comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 4]

11. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞) (T3 vs. R1)
Description: as for outcome 9
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Standard Error); unit: Nanomole*hour/litre (nmol*h/L)
Arm/Group | Cimetidine + R1 (T3) | Cocktail (R1)
Number analyzed (Participants) | 15 | 13
Nanomole*hour/litre (nmol*h/L)
  Furosemide | 202.17 (1.04) | 200.61 (1.05)
  Metformin | 2023.33 (1.06) | 1540.21 (1.07)
  Rosuvastatin | 148.32 (1.13) | 139.21 (1.13)
Statistical Analysis 1: Comparison: Cimetidine + R1 (T3) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean ratio = 100.78, 90% CI 2-sided [93.59 to 108.51], Standard Error of Mean 10.0 — [estimate comment as in outcome 3, analysis 1]; [other analysis details as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Cimetidine + R1 (T3) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 131.37, 90% CI 2-sided [120.37 to 143.37], Standard Error of Mean 13.4 — [estimate comment as in outcome 4, analysis 1]; [other analysis details as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cimetidine + R1 (T3) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 106.55, 90% CI 2-sided [96.87 to 117.19], Standard Error of Mean 12.8 — [estimate comment as in outcome 3, analysis 1]; [other analysis details as in outcome 1, analysis 4]

12. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞) (T4 vs. R1)
Description: as for outcome 9
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Standard Error); unit: Nanomole*hour/litre (nmol*h/L)
Arm/Group | Probenecid + R1 (T4) | Cocktail (R1)
Number analyzed (Participants) | 15 | 16
Nanomole*hour/litre (nmol*h/L)
  Furosemide | 489.28 (1.07) | 188.11 (1.07)
  Metformin | 1346.62 (1.08) | 1330.47 (1.07)
  Rosuvastatin | 244.94 (1.10) | 113.78 (1.10)
Statistical Analysis 1: Comparison: Probenecid + R1 (T4) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean ratio = 260.11, 90% CI 2-sided [237.96 to 284.32], Standard Error of Mean 14.7 — [estimate comment as in outcome 4, analysis 1]; [other analysis details as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Probenecid + R1 (T4) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 101.21, 90% CI 2-sided [95.15 to 107.66], Standard Error of Mean 9.4 — [estimate comment as in outcome 4, analysis 1]; [other analysis details as in outcome 1, analysis 3]
Statistical Analysis 3: Comparison: Probenecid + R1 (T4) vs Cocktail (R1); Test type: Other; ANOVA; Adjusted gMean Ratio = 215.28, 90% CI 2-sided [197.53 to 234.63], Standard Error of Mean 13.1 — [estimate comment as in outcome 4, analysis 1]; [other analysis details as in outcome 1, analysis 4]

ADVERSE EVENTS:
Time Frame: From first drug administration until 7 days thereafter in each treatment period, up to 22 days for part 1 and 27 days for part 2 and 3.
Description: Treatment emergent adverse events (AE's) are presented are on-treatment and treated set (TS) was used for AE reporting.
Groups:
- Rifampin + R1 (T2): Participants were administered a single dose of 600 mg Rifampin film-coated tablet orally with 280 mL of water together with R1 in trial part 1.
- Metformin (R2): Participants were administered a single therapeutic dose of 500 mg Metformin oral solution with 280 mL of water in trial part 2.
- Cimetidine + R1 (T3): Participants were administered 400 mg Cimetidine 1 tablet orally at 1 h prior to R1 and at 4 h, 8 h, 12 h, 24 h (Day 2) and 36 h after R1 (Day 2). All doses of Cimetidine administered with 240 mL water and dose of R1 which is administered with 280 mL of water in trial part 2.
- Cimetidine + R2 (T5): Participants were administered 400 mg Cimetidine 1 tablet orally at 1 h prior to Metformin and at 4 h, 8 h, 12, 24 h (Day 2) and 36 h after therapeutic dose of 500 mg Metformin (Day 2) in trial part 2.
- Furosemide (R3): Participants were administered orally a single therapeutic dose of 40 mg Furosemide oral solution with 280 mL of water in trial part 3.
- Probenecid + R3 (T6): Participants were administered 2 tablets of 500 mg Probenecid (2*500 mg) administered orally 13 hours prior and again 1 h prior to the administration of Furosemide on Day 1 in trial part 3.
Arm/Group | Cocktail (R1) | Verapamil + R1 (T1) | Rifampin + R1 (T2) | Metformin (R2) | Cimetidine + R1 (T3) | Cimetidine + R2 (T5) | Furosemide (R3) | Probenecid + R1 (T4) | Probenecid + R3 (T6)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/12 | 0/12 | 0/16 | 0/17 | 0/17 | 0/16 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/12 | 0/12 | 0/16 | 0/17 | 0/17 | 0/16 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 5/42 | 1/12 | 2/12 | 7/16 | 7/17 | 7/17 | 4/16 | 4/16 | 3/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cocktail (R1) (N=42) | Verapamil + R1 (T1) (N=12) | Rifampin + R1 (T2) (N=12) | Metformin (R2) (N=16) | Cimetidine + R1 (T3) (N=17) | Cimetidine + R2 (T5) (N=17) | Furosemide (R3) (N=16) | Probenecid + R1 (T4) (N=16) | Probenecid + R3 (T6) (N=15)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 1 | 4 | 3 | 2 | 2 | 0 | 1
Orthostatic intolerance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conversion disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT03307252/Prot_001.pdf
  • Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT03307252/SAP_000.pdf